CLINICAL TRIAL: NCT05807581
Title: Clinical, Molecular and Electrophysiological Profiling of Parkinson's Disease: the Role of Non-pharmacological Therapies
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Collaborators: IRCCS National Neurological Institute "C. Mondino" Foundation (Other); Istituto Neurologico Mediterraneo Neuromed S. R. L (Other); Azienda Ospedaliera Universitaria Policlinico "G. Martino" (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 5478
Record Dates: First submitted 2023-03-13; First posted 2023-04-11 (Actual); Last update posted 2024-03-13 (Actual); Status verified 2023-03

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease | interventions — Exercise

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Biomarkers (No Intervention)
- physical activity (Active Comparator)
  Interventions: Other: physical activity
- sedentary (No Intervention)
- iTBS active (Active Comparator)
  Interventions: Other: iTBS
- iTBS sham (Sham Comparator)
  Interventions: Other: iTBS

INTERVENTIONS:
Other: physical activity — treadmill running 3 times weekly
  Arms: physical activity
Other: iTBS — repetitive TMS stimulation 5 days weekly for two weeks
  Arms: iTBS active; iTBS sham

SUMMARY:
In Parkinson's disease (PD), direct evidence linking inflammation to the harmful activities of alpha-synuclein (a-syn) aggregates, the disease onset, and its progression is still lacking. This translational project aims to reveal the causal relationship between a-syn and inflammation. The investigators will also investigate the mechanisms underlying the beneficial effects of two non-pharmacological approaches, motor exercise and neuromodulation, with particular focus on neuroinflammation and brain-derived neurotrophic factor (BDNF) production. the investigators will investigate the molecular pathways and synaptic alterations underlying disease progression. This will be paralleled by a clinical study, in which clinical assessment will be associated with cerebrospinal fluid (CSF) and blood neurodegeneration and inflammatory biomarkers measures. Then, the investigators will test the hypothesis that intensive exercise and neuromodulation may reduce neuroinflammation and a-syn spreading via the activation of BDNF-related pathways.

ELIGIBILITY:
Inclusion Criteria:

* clinically established diagnosis of PD according to the Movement Disorders Society (MDS) diagnostic criteria
* Hoehn & Yahr (H&Y) stage between 1 and 3

Exclusion Criteria:

* Pregnancy
* Oncological or autoimmune comorbidities

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2023-06-09 (Actual); Primary Completion 2025-05-30 (Estimated); Study Completion 2025-05-30 (Estimated)

PRIMARY OUTCOMES:
CLINICAL PROFILING OF PD PATIENTS (n=400) | at enrolling
  patients will be evaluated by means of validated clinical scales Movement disorders society-unified Parkinson's Disease Rating Scale (min 0- max 260, better clinical conditions has lower scores)
CLINICAL PROFILING OF PD PATIENTS (n=400) | at enrolling
  patients will be evaluated by means of validated clinical scales Non-Motor Symptoms scale (min 0- 360 max , better clinical conditions has lower scores)
MOLECULAR PROFILING OF PD PATIENTS (n=400) | at enrolling
  Biomarkers related to axonal damage (total tau (t-Tau), neurofilament light chain, (NfL), and phosphorylated neurofilament heavy chain, (p-NfH), synaptic dysfunction (a-synuclein (a-syn) and neurogranin, (Ng)), neuroinflammation (soluble triggering receptor expressed on myeloid cells 2, sTREM2, and chitinase-3- like protein 1, YKL-40) will be analysed in cerebrospinal fluid (CSF) and blood samples and extracellular vesicles (EVs) (UO1, UO2) (for all the biomarkers, ng/ml).
ELECTROPHYSIOLOGICAL PROFILING OF PD PATIENTS (n=400) | at enrolling
  Motor evoked potentials (MEPs) from the First Digital Interosseus muscle of the most affected hand of each patient, a brief pattern of iTBS will be applied to promote enhancement of cortical excitability. MEPs size will be then assessed again using single-pulse TMS.

SECONDARY OUTCOMES:
UPDRS CHANGES AFTER NON-PHARMACOLOGICAL INTERVENTIONS (n=240) CLINICAL PROFILING OF PD PATIENTS (n=400) | at the end of the non-pharmacological intervention (2 weeks for TMS branches, 3 months for physical activity branches) and 3 and 6 months after
  patients will be evaluated by means of validated clinical scales, Movement disorders society- Unified Parkinson's disease rating scale, (min 0- 260 max , better clinical conditions has lower scores)
NMSS CHANGES AFTER NON-PHARMACOLOGICAL INTERVENTIONS (n=240) CLINICAL PROFILING OF PD PATIENTS (n=400) | at the end of the non-pharmacological intervention (2 weeks for TMS branches, 3 months for physical activity branches) and 3 and 6 months after
  patients will be evaluated by means of validated clinical scales Non-Motor Symptoms Scale (min 0- 360 max , better clinical conditions has lower scores)
MOLECULAR CHANGES AFTER NON-PHARMACOLOGICAL INTERVENTIONS (n=240) | at the end of the non-pharmacological intervention (2 weeks for TMS branches, 3 months for physical activity branches) and 3 and 6 months after
  Biomarkers related to axonal damage (total tau (t-Tau), neurofilament light chain, (NfL), and phosphorylated neurofilament heavy chain, (p-NfH), synaptic dysfunction (a-synuclein (a-syn) and neurogranin, (Ng)), neuroinflammation (soluble triggering receptor expressed on myeloid cells 2, sTREM2, and chitinase-3- like protein 1, YKL-40) will be analysed in cerebrospinal fluid (CSF) and blood samples and extracellular vesicles (EVs) (UO1, UO2) (for all the biomarkers, ng/ml).
ELECTROPHYSIOLOGICAL CHANGES AFTER NON-PHARMACOLOGICAL INTERVENTIONS (n=240) | at the end of the non-pharmacological intervention (2 weeks for TMS branches, 3 months for physical activity branches) and 3 and 6 months after
  Motor evoked potentials (MEPs) from the FDI muscle of the most affected hand of each patient, a brief pattern of iTBS will be applied to promote enhancement of cortical excitability. MEPs size will be then assessed again using single-pulse TMS.

CONTACTS AND LOCATIONS:
Locations (1):
- Fondazione Policlinico Universitario Agostino Gemelli IRCCS, Roma, Italy

IPD SHARING:
Plan to Share IPD: No